CLINICAL TRIAL: NCT03512756
Title: A Randomized Phase 2/3 Multi-Center Study of SM-88 in Subjects With Pancreatic Cancer Whose Disease Has Progressed or Recurred
Brief Title: A Randomized Phase 2/3 Multi-Center Study of SM-88 in Participants With Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Tyme, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Tyme-88-Panc
Record Dates: First submitted 2018-04-18; First posted 2018-05-01 (Actual); Results first posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Pancreas cancer; Pancreatic; Pancreas; cancer; low toxicity; chemotherapy; metastatic; SM-88; SM88; 3rd line; third line; CMBT; well tolerated; MPS; Racemetyrosine; Methoxsalen; Sirolimus; Phenytoin
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Methoxsalen; Phenytoin; Sirolimus; racemetyrosine; Capecitabine; Gemcitabine; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 and Part 2 SM-88 Arm (Experimental): (Part 1 enrollment complete) SM-88 used with MPS (methoxsalen, phenytoin and sirolimus)
  (Part 2 actively enrolling) SM-88 (920 mg per day) used with MPS (methoxsalen, phenytoin and sirolimus) will be administered to 125 evaluable participants until unacceptable toxicity, disease progression, or any of the treatment discontinuation criteria are met.
  Interventions: Drug: SM-88 used with MPS (methoxsalen, phenytoin, sirolimus)
- Physician's Choice (Experimental): Physician's Choice therapy will be administered for a total of 125 evaluable participants until unacceptable toxicity, disease progression, or any of the treatment discontinuation criteria are met.
  Interventions: Drug: Capecitabine, Gemcitabine, and 5-FU

INTERVENTIONS:
Drug: SM-88 used with MPS (methoxsalen, phenytoin, sirolimus) — Daily oral therapy for cancer
  Other Names: SM-88; Racemetyrosine
  Arms: Part 1 and Part 2 SM-88 Arm
Drug: Capecitabine, Gemcitabine, and 5-FU — Investigator choice of the following therapies:
  Capecitabine, Gemcitabine, and 5-FU
  Other Names: Physician's Choice
  Arms: Physician's Choice

SUMMARY:
A prospective, open-label phase 2/3 trial in metastatic pancreatic cancer participants who have failed two lines of prior systemic therapy. The trial is designed to evaluate the safety and efficacy of SM-88 used with MPS (methoxsalen, phenytoin and sirolimus) in pancreatic cancer and will measure multiple endpoints, including overall survival, progression free survival, relevant biomarkers, quality of life, safety, and overall response rate.

(Part 1 enrollment complete) In the initial stage of the trial (36 participants), two dose levels of SM-88's metyrosine-derivative was evaluated.

(Part 2 actively enrolling) The second part will consist of a subsequent expansion of the trial to further assess safety and efficacy of SM-88 used with MPS containing the selected SM-88 RP2D from Part 1. A total of 250 participants in the second part will be randomized 1:1 either to the SM-88 arm (125 participants) or Physician's Choice of therapy for the Control Arm (125 participants). Participants should have previously received two lines of prior systemic therapy.

DETAILED DESCRIPTION:
Please refer to Inclusion/Exclusion Criteria and Summary

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1.

Part 1

Biopsy-proven metastatic pancreatic adenocarcinoma with documented radiographic disease progression on or after one or more systemic therapies. Chemotherapy given as part of prior chemoradiation in the setting of non-metastatic pancreatic cancer does not count as a line of therapy. Chemotherapy given for at least 4 months as adjuvant after complete response is considered as a first line therapy.

Part 2

Biopsy-proven metastatic pancreatic adenocarcinoma on or after two prior lines of systemic therapy. Chemotherapy given as part of prior chemo- radiation in the setting of non-metastatic pancreatic cancer does not count as a line of therapy unless metastases develop within 6 months of completing the chemo sensitization. Chemotherapy given for at least 4 months as adjuvant after a CR to any therapy (e.g. surgery and radiation therapy) is also considered as a first line therapy. Of the two prior lines, participants should have received a gemcitabine-based regimen for a prior line and a 5-FU based regimen as a prior line of therapy. Investigational therapies as part of a prior line regimen are permitted.

2. Participants Have received two (2) and not more than two (2) previous systemic regimens for the treatment of pancreatic adenocarcinoma

3. Must be eligible to receive one or more of the Physician Choice options.

4. Radiographically measurable disease of at least one site by CT scan (or MRI, if allergic to CT contrast media). Imaging results must be obtained within the 14-day window prior to randomization

5. Must have completed any investigational cancer therapy at least 30 days prior to first dose.

6. Must have completed any other cancer therapy at least 14 days prior to first dose and recovered from major side effects of prior therapies or procedures.

7. ≥18 years of age.

8. ECOG PS ≤2.

9. Adequate organ function defined as follows (lab results must be obtained within the 7-day window prior to randomization):

1. All laboratory parameters ≤ Grade 2 NCI Common Terminology Criteria for Adverse Events (CTCAE) criteria.
2. In addition:

i. Hematologic: Platelets ≥ 100 x 109 g/dL; Absolute Neutrophil Count ≥ 1.5 x 109/L (without platelet transfusion or growth factors within the 7 days prior to the screening laboratory assessment).

ii. Hepatic: transaminase /alanine transaminase ≤ 2.5 x upper limit of normal (ULN); total or conjugated bilirubin ≤ 1.5 x ULN, alkaline phosphatase (ALP) < 2.5 x ULN.

iii. Renal: serum creatinine ≤1.5 x ULN and creatinine clearance ≥ 60 mL/min as calculated by the Cockroft-Gault method.

iv. Coagulation: International normalized ratio (INR) ≤ 1.2 within 28 days of starting study.

v. Albumin: ≥ 3.0 g/dL. vi. Weight: No more than a 5% change from Screening to Randomization (must be at least 1 week apart).

10. All acute toxic effects of any prior antitumor therapy resolved to Grade ≤ 1 before baseline, with the exception of alopecia and neurotoxicity (CTCAE Grade 1 or 2 permitted).

11. Able and willing to provide written informed consent to participate in this study.

12.Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

13. Must be able to swallow whole capsules.

14. Females must either be of non-reproductive potential, not breast-feeding or must have a negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on Day 1.

15. Participant of fertile potential who engage in heterosexual intercourse with partners of childbearing potential must attest to the use of highly effective contraception while enrolled in the study and for at least 6 months following the last dose of study drug.

Highly effective birth control methods include the following (the participantshould choose 2 to be used with their partner):

1. Oral, injectable, or implanted hormonal contraceptives.
2. Condom with a spermicidal foam, gel, film, cream, or suppository.
3. Occlusive cap (diaphragm or cervical/vault cap) with a spermicidal foam, gel, film, cream, or suppository.

Or any one of the following:

1. Intrauterine device.
2. Intrauterine system (for example, progestin-releasing coil).
3. Vasectomized male (as determined by the investigator).
4. Tubal ligation/sterilization (female).

Exclusion criteria for Parts 1 and 2 are as follows:

1. Any screening laboratory, ECG, or other findings that, in the opinion of the investigator, medical monitor or the sponsor, indicate an unacceptable risk for the participant's participation in the study.
2. History or evidence of any clinically significant disorder, condition, or disease that, in the opinion of the investigator or medical monitor would pose a risk to the participant's safety or interfere with the study evaluations, procedures, or completion. Examples include intercurrent illness such as active uncontrolled infection, active or chronic bleeding event within 28 days of baseline, uncontrolled cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.
3. History of a concurrent or second malignancy, except for adequately treated localized basal cell or squamous cell carcinoma of the skin, adequately treated superficial bladder cancer, adequately treated Stage 1 or 2 cancer currently in complete remission; or any other cancer that has been in complete remission for ≥ 5 years.
4. Participants with MSI-H pancreatic cancer who have not previously received pembrolizumab.
5. Any known actionable mutation (e.g. BRCA mutation) who have not been treated with an approved drug for the mutation (the drug does not have to be approved for the indication).
6. Radiation to all target lesions within 12 weeks of study baseline.
7. No measurable target lesions.
8. Current use, or up to 14 days prior use, of a restricted medication (see Section 8.7) or requires any of these medications during treatment phase.
9. Major surgery, defined as any surgical procedure that involves general anesthesia and a significant incision (i.e. larger than that required for placement of central venous access, percutaneous feeding tube, or biopsy) within 28 days of the first dose of study drug.
10. Minor surgical procedures within 7 days of baseline, or not yet recovered from any prior surgery.
11. Any dysphagia, odynophagia, esophageal dysmotility or stricture, known gastrointestinal (GI) malabsorption syndrome, or intractable diarrhea that may significantly alter the absorption of any of the components of SM-88 used with MPS, e.g., cirrhosis.
12. Known human immunodeficiency (HIV) virus infection. Note: HIV testing is not required in the absence of clinical suspicion.
13. Known hepatitis B surface antigen (HBsAg) positive.
14. Known hepatitis C (HCV) viral RNA present.
15. Have previously been enrolled in this study or any other study investigating SM-88 or who have previously received any SM-88, methoxsalen, phenytoin, or sirolimus in a clinical trial.
16. History of any known drug allergies to any study medication.
17. Are currently enrolled in, or have discontinued within 14 days of screening, from a clinical trial involving an investigational product or non-approved use of a drug or device.
18. Must not have any clinically significant and uncontrolled major medical condition(s) including, but not limited to uncontrolled nausea/vomiting/diarrhea; active uncontrolled infection; symptomatic congestive heart failure (New York Heart Association [NYHA] class ≥ II); unstable angina pectoris or cardiac arrhythmia; psychiatric illness/social situation that would limit compliance with study requirements.
19. >5% weight loss over the 28 days prior to consent or >5% change in weight from consent to randomization.
20. Participants that have a variety of factors influencing oral drugs (such as unable to swallow, nausea, vomiting, chronic diarrhea and intestinal obstruction, etc.).
21. Central nervous system metastasis; with the exception of participants who have stable brain metastases as defined as off steroids and no CNS progress for 6 months after CNS treatment.
22. Pregnant or lactating women.
23. Substance abuse that cannot be ended, or participants with mental disorders that will prevent compliance or evaluation including uncontrolled schizophrenia, uncontrolled depression or other uncontrolled disorders.
24. History of hypersensitivity to phenytoin, its inactive ingredients, or other hydantoins; or a history of prior acute hepatotoxicity attributable to phenytoin.
25. Participants exhibiting idiosyncratic reactions to psoralen compounds.
26. Participants with a hypersensitivity to sirolimus.
27. Participants with a history of the light sensitive diseases for which methoxsalen would be contraindicated. Diseases associated with photosensitivity include lupus erythematosus, porphyria cutanea tarda, erythropoietic protoporphyria, variegate porphyria, xeroderma pigmentosum, and albinism.
28. Participants treated, or anticipated to be treated, with delavirdine (due to potential for loss of virologic response and possible resistance to delavirdine or to the class of non-nucleoside reverse transcriptase inhibitors caused by phenytoin).
29. Participants with cutaneous melanoma or invasive squamous cell carcinomas or a history thereof, except for those in complete remission for ≥5 years (due to contraindication for use of methoxsalen).
30. Participants with prior organ transplant or being treated, or anticipated to be treated, with cyclosporine (because long-term administration of the combination of cyclosporine and sirolimus is associated with deterioration of renal function).
31. Participants with a seizure disorder that is not well controlled or who have required a change in seizure medications within 60 days of enrollment to the trial.
32. Participants treated, or anticipated to be treated, with a calcineurin inhibitor (because concomitant use of sirolimus and a calcineurin inhibitor increases the risk of calcineurin inhibitor-induced hemolytic uremic syndrome/thrombotic thrombocytopenic purpura/thrombotic microangiopathy [HUS/TTP/TMA]).
33. Participants with interstitial lung disease (ILD) [including pneumonitis, bronchiolitis obliterans organizing pneumonia (BOOP), and pulmonary fibrosis].
34. Baseline repeated prolongation of QT/QTc interval [e.g. > 480 milliseconds (ms)] (CTCAE Grade 1) using Fredericia's QT correction formula.
35. A family history of Long QT Syndrome or Torsades de Pointes
36. Clinically significant cataracts or aphakia.
37. Presence of ascites or pleural effusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe DelPriore, MD, MPH, Study Director — Tyme, Inc
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City Of Hope, Duarte, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Hartford Healthcare Cancer, New Britain, Connecticut
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Advent Health Florida Hospital Tampa, Tampa, Florida
  - June E. Nylen Cancer Center, Sioux City, Iowa
  - University Medical Center, New Orleans, Louisiana
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - North Shore Hematology Oncology, East Setauket, New York
  - NY Cancer and Blood Specialist, East Setauket, New York
  - NYU Langone Health, New York, New York
  - Central Park Hematology & Oncology, New York, New York
  - Weill Cornell, New York, New York
  - New York Cancer and Blood Specialist, The Bronx, New York
  - The Ohio State University, Columbus, Ohio
  - Texas Oncology-Baylor, Dallas, Texas
  - MD Anderson, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noel MS, Kim S, Hartley ML, Wong S, Picozzi VJ, Staszewski H, Kim DW, Van Tornout JM, Philip PA, Chung V, Ocean AJ, Wang-Gillam A. A randomized phase II study of SM-88 plus methoxsalen, phenytoin, and sirolimus in patients with metastatic pancreatic cancer treated in the second line and beyond. Cancer Med. 2022 Nov;11(22):4169-4181. doi: 10.1002/cam4.4768. Epub 2022 May 2. PMID 35499204

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a two-part study.
  The first part (Part 1) was used to determine which dose of SM-88 was to be selected for further study (recommended for Phase 2 dose [RP2D]).
  The second part (Part 2) consisted of an expansion cohort of participants at the selected dose of Physician's Choice therapies.
Groups:
- Part 1: SM-88 460 Milligrams (mg): Participants received 230 mg SM-88 oral tablets twice daily along with methoxsalen, phenytoin, and sirolimus (MPS) for up to 6 months
- Part 1: SM-88 920 mg; Part 2: SM-88 920 mg: Participants received 460 mg SM-88 oral tablets twice daily along with MPS for up to 6 months
- Part 2: Physician's Choice: Participants received one of capecitabine, gemcitabine or 5-fluorouracil (FU) per the physician's choice
Period: Part 1
Arm/Group | Part 1: SM-88 460 Milligrams (mg) | Part 1: SM-88 920 mg | Part 2: SM-88 920 mg | Part 2: Physician's Choice
Started | 25 | 24 | 0 (No participants were enrolled in this arm during Part 1.) | 0 (No participants were enrolled in this arm during Part 1.)
Received At Least 1 Dose of Study Drug (Per protocol, only participants in this row have been included in the Safety Analysis Population, and have been used to report Baseline Measures and Adverse Events.) | 25 | 23 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 25 | 24 | 0 | 0
Not completed — Death | 23 | 18 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0
Period: Part 2
Arm/Group | Part 1: SM-88 460 Milligrams (mg) | Part 1: SM-88 920 mg | Part 2: SM-88 920 mg | Part 2: Physician's Choice
Started | 0 (No participants were enrolled in this arm during Part 2.) | 0 (No participants were enrolled in this arm during Part 2.) | 41 | 40
Received At Least 1 Dose of Study Drug (Per protocol, only participants in this row have been included in the Safety Analysis Population, and have been used to report Baseline Measures and Adverse Events.) | 0 | 0 | 40 | 30
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 41 | 40
Not completed — Death | 0 | 0 | 32 | 21
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 4
Not completed — Study Terminated by Sponsor | 0 | 0 | 2 | 6
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 9

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants enrolled in the study who received at least one dose of study drug, and assigned to treatment actually received.
Groups:
- Part 1: SM-88 460 mg: Participants received 230 mg SM-88 oral tablets twice daily along with MPS for up to 6 months
- Part 2: Physician's Choice: Participants received one of capecitabine, gemcitabine or 5-FU per the physician's choice
- Total: Total of all reporting groups
Arm/Group | Part 1: SM-88 460 mg | Part 1: SM-88 920 mg | Part 2: SM-88 920 mg | Part 2: Physician's Choice | Total
Number analyzed (Participants) | 25 | 23 | 40 | 30 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22 | 7 | 51
  >=65 years | 14 | 12 | 18 | 23 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 14 | 13 | 50
  Male | 14 | 11 | 26 | 17 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 7 | 1 | 9
  Not Hispanic or Latino | 24 | 23 | 33 | 29 | 109
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3 | 6
  White | 25 | 21 | 33 | 19 | 98
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the number of days between the first study drug administration and death from any cause. Results are reported in weeks.
Time Frame: Up to 12 months
Population: Evaluable Population included all participants enrolled in the study who received at least 1 cycle (28 days) of study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this Outcome Measure.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Part 1: SM-88 460 mg | Part 1: SM-88 920 mg | Part 2: SM-88 920 mg | Part 2: Physician's Choice
Number analyzed (Participants) | 20 | 17 | 33 | 27
Weeks | 21.3 [9.7 to 35.0] | 15.7 [11.1 to 24.7] | 14.0 [11.1 to 19.4] | 24.1 [13.7 to 31.6]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-Free Survival (PFS), is defined as the time from randomization to first documentation of objective tumor progression (progressive disease) or death due to any reasons whichever comes first. Disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Results are reported in weeks.
Time Frame: Up to 12 months
Population: Intent to Treat (ITT) Population included all participants who consented in the study and randomized to treatment, and assigned to treatment they were randomized to. Here, 'Overall number of participants analyzed' = participants evaluable for this Outcome Measure.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Part 1: SM-88 460 mg | Part 1: SM-88 920 mg | Part 2: SM-88 920 mg | Part 2: Physician's Choice
Number analyzed (Participants) | 25 | 24 | 41 | 40
Weeks | 8.0 [7.1 to 8.6] | 8.0 [5.6 to 11.1] | 7.7 [5.6 to 8.0] | 8.9 [6.0 to 12.7]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality are reported from participant randomization up to 12 months. Serious and Other Adverse Events are reported from the date of first dose to 28 days after the date of last dose (up to 12 months)
Description: All-cause mortality was assessed in all enrolled participants.
  Safety Analysis Population was used to report Serious and Other Adverse Events. It included all participants enrolled in the study who received at least one dose of study drug, and assigned to treatment actually received.
Arm/Group | Part 1: SM-88 460 mg | Part 1: SM-88 920 mg | Part 2: SM-88 920 mg | Part 2: Physician's Choice
All-Cause Mortality (participants affected / at risk) | 23/25 | 18/24 | 32/41 | 21/40
Serious Adverse Events (participants affected / at risk) | 14/25 | 12/23 | 19/40 | 11/30
Other Adverse Events (participants affected / at risk) | 12/25 | 10/23 | 23/40 | 18/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: SM-88 460 mg (N=25) | Part 1: SM-88 920 mg (N=23) | Part 2: SM-88 920 mg (N=40) | Part 2: Physician's Choice (N=30)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 5 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 3 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0 | 0
Afferent loop syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 2 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: SM-88 460 mg (N=25) | Part 1: SM-88 920 mg (N=23) | Part 2: SM-88 920 mg (N=40) | Part 2: Physician's Choice (N=30)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 4 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Systemic candida (Infections and infestations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 3 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 3
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Depression (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Embolic stroke (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT03512756/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT03512756/SAP_001.pdf